CLINICAL TRIAL: NCT05580497
Title: Soft Robotics for Improved Standing and Walking in Infants With Cerebral Palsy
Brief Title: Soft Robotics for Infants With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor and Chairman, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021.171
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soft Wearable Robotic Knee System (Experimental): 30 minutes gait training wearing the Soft Wearable Robotic Knee System
  Interventions: Device: Soft Wearable Robotic Knee System

INTERVENTIONS:
Device: Soft Wearable Robotic Knee System — Power assistance will be provided from the motor to the knee joint

SUMMARY:
Children with spastic cerebral palsy suffer from significant weakness that contributes to abnormal posture and movement. It is thought that this arises due lack of frequency sufficient tension to encourage normal muscular growth underlying the need for early intervention to encourage walking. The failure of muscle growth to keep pace with bone growth is most evident in the bi-articular muscles and contributes to joint contractures and gait abnormalities such as toe-walking and flexed-knee gait.

Recently, our research team has developed a novel, lightweight (0.2kg at knee joint) and portable (energetically autonomous) Soft Wearable Robotic Knee System that can provide active powered knee assistance and synchronized proprioceptive feedback for the gait training of stroke patients' standing and walking.

ELIGIBILITY:
Inclusion Criteria:

* capable of understanding the proposed exercises;
* aged 2 to 15 years;
* maximum weight 75 kg;
* children with no deformations that could prevent the use of the exoskeleton;
* Gross Motor Function Classification System (GMFCS) levels I to III;
* able to signal pain or discomfort.

Exclusion Criteria:

* unhealed skin lesions in the lower limbs;
* aggressive or self-harming behaviors;
* severe cognitive impairment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Classification System | Within one month after the last training session
  It categorized the gross motor function of children and young people with cerebral palsy into 5 different levels. With level 1: Children walk at home, school, outdoors and in the community, while level 5: Children are transported in a manual wheelchair in all settings.

SECONDARY OUTCOMES:
6-Minute-Walk Test | Within one month after the last training session
  It is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
10-Meter-Walk Test | Within one month after the last training session
  It is a performance measure used to assess walking speed in meters per second over a short distance.
Timed Up and Go test | Within one month after the last training session
  It is used to determine fall risk and measure the progress of balance, sit to stand and walking.
Five Times Sit to Stand Test | Within one month after the last training session
  It is used to assess functional lower extremity strength, transitional movements, balance, and fall risk.
Berg Balance Scale | Within one month after the last training session
  It is used to objectively determine a person's ability to safely balance during a series of predetermined tasks. It is a 14-item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Department of Biomedical Engineering, The Chinese University of Hong Kong
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No